CLINICAL TRIAL: NCT03249532
Title: Effect of High-volume Online hemodiafiLtration on Intra-diaLytic hemodynAmic (iN)sTability and Cardiac Function in Chronic Hemodialysis Patients (the HOLLANT Study)
Brief Title: Effect of Dialysis Techniques on Blood Pressure and Cardiac Function During Dialysis
Acronym: HOLLANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Niercentrum aan de Amstel, Amstelveen, Netherlands (Unknown); B.Braun Avitum AG (Industry)
Responsible Party: Principal Investigator, M.P.C. Grooteman, MD PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ABR 61210
Record Dates: First submitted 2017-05-23; First posted 2017-08-15 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: End Stage Renal Disease (ESRD); Hemodialysis; Hemodiafiltration; Intradialytic Hypotension; Diastolic Dysfunction
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: prospective, cross over, randomized order
Who Masked: Outcomes Assessor
Masking Description: treatment period will not be available to the assessors of secondary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- standard hemodialysis (Active Comparator): prescription of dialysate temperature: 36.5 degrees celsius prescription of convection volume: 0 Liters (L)
  Interventions: Device: cool hemodialysis; Device: low volume hemodiafiltration; Device: high volume hemodiafiltration
- cool hemodialysis (Active Comparator): prescription of dialysate temperature: 35.5 degrees celsius prescription of convection volume: 0 L
  Interventions: Device: standard hemodialysis; Device: low volume hemodiafiltration; Device: high volume hemodiafiltration
- low volume hemodiafiltration (Active Comparator): prescription of dialysate temperature: 36.5 degrees celsius prescription of convection volume: 15 L
  Interventions: Device: standard hemodialysis; Device: cool hemodialysis; Device: high volume hemodiafiltration
- high volume hemodiafiltration (Active Comparator): prescription of dialysate temperature: 36.5 degrees celsius prescription of convection volume: 25 L
  Interventions: Device: standard hemodialysis; Device: cool hemodialysis; Device: low volume hemodiafiltration

INTERVENTIONS:
Device: standard hemodialysis — hemodialysis with high-flux dialyzer; prescription of dialysate temperature: 36.5 degrees Celsius; convection volume: not applicable
  Arms: cool hemodialysis; high volume hemodiafiltration; low volume hemodiafiltration
Device: cool hemodialysis — hemodialysis with high-flux dialyzer; prescription of dialysate temperature: 35.5 degrees Celsius; convection volume: not applicable
  Arms: high volume hemodiafiltration; low volume hemodiafiltration; standard hemodialysis
Device: low volume hemodiafiltration — hemodiafiltration; prescription of dialysate temperature: 36.5 degrees celsius prescription of convection volume: 15 L
  Arms: cool hemodialysis; high volume hemodiafiltration; standard hemodialysis
Device: high volume hemodiafiltration — hemodiafiltration; prescription of dialysate temperature: 36.5 degrees celsius prescription of convection volume: 25 L
  Arms: cool hemodialysis; low volume hemodiafiltration; standard hemodialysis

SUMMARY:
Online hemodiafiltration confers a reduced mortality risk. However, it is not clear why HDF improved survival. To gain more insight in this issue, the effect of 4 dialysis techniques (differing in dialysate temperature and the absence/presence of convective clearance) on intradialytic hemodynamic stability and cardiac function will be investigated in a prospective cross over trial.

DETAILED DESCRIPTION:
Despite the use of high permeable dialyzers, which combine diffusive with convective clearance, the clinical outcome of hemodialysis (HD) patients remains poor. In post-dilution online hemodiafiltration (denoted further on as HDF) diffusive clearance is similar to HD, while the amount of convective transport is considerable increased. Recently, 4 randomized controlled trails have been published which compared HD with HDF. Although the results of the individual studies were inconclusive, a recent meta-analysis, using individual patient data of these studies, showed a superior outcome for patients treated with HDF. The largest mortality reduction was obtained in patients receiving the highest convection volume (high-volume HDF [HV-HDF] >23 L/1.73 m2/session): all-cause mortality [22% (95 % confidence interval [CI] 2-38)], cardiovascular disease (CVD) mortality [31% (95 % CI 0-53)].

It is far from clear, however, why (HV)HDF is associated with an improved survival. Both long term and short term effects may be involved. With respect to the latter, the intra-dialytic removal of middle molecular weight (MMW) uremic retention products and a superior bio-incompatibility (BI) profile may play a role. In addition, treatment with HDF may induce less intra-dialytic hypotension (IDH) and less tissue injury. Enhanced removal of the MMW substance FGF23 may reduce the intra-dialytic acute phase reaction (APR), which is regarded a chief element of HD-induced BI. Other key components which may contribute to IDH and are supposed to be alleviated by HDF, include dialysis-induced hypoxia and intra-dialytic extracellular vesicle release. Patho-physiologically, IDH depends both on a decline in the circulating blood volume and an impaired response to hypovolaemia. As a result, venous return, cardiac output and peripheral vascular resistance are impaired. Since IDH is reduced by HD with cool dialysate (C-HD), thermal factors may play an important role.

Microcirculatory dysfunction is a prominent feature of HD patients. Since IDH occurs in 20-30% of the sessions, any interference with an already abnormal perfusion may further deteriorate the structure and function of vital organs, such as the brain, gut and heart. HD-associated cardiomyopathy, which is considered a model of repetitive organ ischemia-reperfusion injury, is superimposed on the cardiac changes resulting from the various inflammatory and metabolic derangements of pre-dialysis kidney disease. As measured by imaging techniques and biomarkers, HD induces a fall in cardiac perfusion and elicits tissue injury. While cardiac MRI is considered the reference method for LV quantification, intra-dialytic measurements can only be obtained in stable patients who can be safely transferred to the radiology department. Echocardiography, though, can be performed in all individuals at the bed-side, including hypotension-prone patients. Because of its superiority over standard echocardiography, especially with respect to diastolic (dys)function, speckle tracking echocardiography will be used in the present study.

As mentioned, the effect on long term survival is especially prominent when HV-HDF is applied. Theoretically, HV-HDF is also the preferred treatment to circumvent dialysis-induced IDH, and hence, to alleviate the repetitive intra-dialytic tissue damage. Therefore, the following hypotheses will be tested:

1. intra-dialytic hemodynamic stability is better preserved during HV-HDF as compared to standard (S)-HD, C-HD and low volume (LV)-HDF;
2. mainly as a result of a better intra-dialytic hemodynamic stability, the severity of organ injury, especially the heart, is least evident during HV-HDF;
3. the mechanism of a better preserved intra-dialytic hemodynamic stability during HV-HDF depends on its superior thermal balance and/or bio-incompatibility, clearance of MMW substances, or a combination of these items.

Worldwide, however, (HV)HDF is only limited available. Since intradialytic hemodynamic instability may contribute substantially to the poor clinical prospects of end-stage-kidney-disease (ESKD) patients, these individuals may benefit from each maneuver that minimizes the number and severity of intradialytic hypotensive episodes. Therefore, the question which of the comparator treatments [(S)-HD, C-HD and LV-HDF] has the best intradialytic hemodynamic stability, appears relevant as well.

ELIGIBILITY:
Inclusion Criteria:

* treatment with HD or HDF 3 x per week during at least 4 hours for at least 2 months
* ability to understand study procedures
* willingness to provide informed consent
* single pool Kt/V urea (spKt/Vurea) ≥ 1.2
* achievement of blood flow of ≥360 ml/min and/or convection volume of >23 Liter per treatment during the run-in phase

Exclusion Criteria:

* - current age < 18 years
* severe incompliance to dialysis procedure and accompanying prescriptions, especially frequency and duration of dialysis treatment
* life expectancy < 3 months
* participation in another clinical intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
intradialytic hypotension | up to 4 hours (= one dialysis treatment); assessed during 3 treatments on each modality
  nadir in systolic blood pressure (SBP) of 90 mmHg for patient with predialysis SBP <160mmHg and a nadir of 100 mmHg for patients with predialysis SBP ≥160 mmHg during treatment (blood pressure will be measured before and every 15 minutes after the start of dialysis during the treatment)

SECONDARY OUTCOMES:
diastolic dysfunction during treatment | up to 4 hours (= one dialysis treatment); assessed during 1 treatment on each modality
  speckle tracking echocardiography will be performed before, after 60 minutes of dialysis and after and after 3,5 hours

OTHER OUTCOMES:
systolic blood pressure | up to 4 hours(= one dialysis treatment); assessed during 3 treatments on each modality
  change in systolic blood pressure (mmHg)
diastolic blood pressure | up to 4 hours(= one dialysis treatment); assessed during 3 treatments on each modality
  change in diastolic blood pressure (mmHg)
mean arterial blood pressure | up to 4 hours(= one dialysis treatment); assessed during 3 treatments on each modality
  change in mean arterial blood pressure (mmHg)
pulse pressure | up to 4 hours(= one dialysis treatment); assessed during 3 treatments on each modality
  change in pulse pressure (systolic - diastolic blood pressure; mmHg)
beat-to-beat blood pressure | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  change in beat-to-beat blood pressure (finger cuff; mmHg)
heart rate | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  change in heart rate (finger cuff assessment)
stroke volume | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  change in stroke volume (finger cuff assessment)
cardiac output | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  change in cardiac output (finger cuff assessment)
total peripheral resistance | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  change in total peripheral resistance (finger cuff assessment)
number of sessions with reached target dry weight | up to 4 hours(= one dialysis treatment); assessed during 3 treatments on each modality
  number of sessions with reached target dry weight (kg)
relative blood volume | up to 4 hours(= one dialysis treatment); assessed during 2 treatments on each modality
  relative blood volume (%) during dialysis treatment
oxygen saturation | up to 4 hours(= one dialysis treatment); assessed during 2 treatments on each modality
  oxygen saturation in the arterial line of the extracorporeal system (%) during dialysis treatment; patients with central venous catheters and fistulas/grafts will be analyzed separately
oxygen partial pressure (pO2) | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  pO2 in the arterial line of the extracorporeal system (mmHg or kiloPascal [kPa], assessed by a point of care device) during dialysis treatment; patients with central venous catheters and fistulas/grafts will be analyzed separately
change in creatine kinase (CK)-MB | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of cardiac damage, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment
change in bacterial DNA in blood | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of gut ischemia, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment
change in soluble CD14 | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of gut ischemia, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment
change in extracellular vesicles (EVs) | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of endothelial damage, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment
change in soluble intercellular adhesion molecule-1 (s-ICAM-1) | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of endothelial damage, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment
change in high sensitivity C-reactive protein (hs-CRP) | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of inflammation, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment
change in interleukin-6 (IL-6) | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of inflammation, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment
change in fibroblast growth factor-23 (FGF-23) | up to 4 hours(= one dialysis treatment); assessed during 1 treatment on each modality
  marker of inflammation/mineral bone disease, assessment in blood from arterial line of extracorporeal circuit, before and after dialysis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Muriel PC Grooteman, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (3):
- Netherlands (3):
  - St Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Niercentrum aan de Amstel, Amstelveen
  - VUmc, Amsterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rootjes PA, Nube MJ, de Roij van Zuijdewijn CLM, Wijngaarden G, Grooteman MPC. Effect of various dialysis modalities on intradialytic hemodynamics, tissue injury and patient discomfort in chronic dialysis patients: design of a randomized cross-over study (HOLLANT). BMC Nephrol. 2021 Apr 15;22(1):131. doi: 10.1186/s12882-021-02331-z. PMID 33858390